CLINICAL TRIAL: NCT00103311
Title: A Randomized Phase II Non-Comparative Study of SB-715992 Given Weekly or Every Three Weeks in Advanced or Metastatic Colorectal Cancer
Brief Title: SB-715992 in Treating Patients With Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02834; NCI-2012-02834 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-51 (Other: City of Hope); 6800 (Other: CTEP)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2013-10

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IIIA Colon Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — ispinesib

ARMS (2):
- Arm I (Experimental): Patients receive SB-715992 IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ispinesib; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients receive SB-715992 IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ispinesib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: ispinesib — Given IV
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well SB-715992 works in treating patients with advanced or metastatic colorectal cancer. Drugs used in chemotherapy, such as SB-715992, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate in patients with advanced or metastatic colorectal cancer treated with SB-715992 once a week for 3 weeks, every 28 days and SB-715992 once every 21 days.

SECONDARY OBJECTIVES:

I. To determine the time to tumor progression, progression free and overall survival of patients and toxicity in patients with advanced or metastatic colorectal cancer treated with SB-715992 once a week for 3 weeks, every 28 days and SB-715992 once every 21 days.

II. To characterize the population pharmacokinetic (PK) parameters of SB-715992 including an assessment of significant covariates on SB-715992 PK and an assessment of the potential relationships between the pharmacokinetics of SB-715992 and relevant safety and efficacy endpoints.

IV. To examine cytoskeletal morphology changes in response to SB-715992 in peripheral blood mononuclear cells and tumors by fluorescent immunohistochemistry.

V. To evaluate mRNA expression of betaΙΙΙ-tubulin and KSP in archival tumor tissue.

VI. To determine the frequency of genomic polymorphisms in genes targeted by SB-715992 (measured in peripheral blood mononuclear cells) and to assess whether germline polymorphisms (DNA) of genes targeted by SB-715992 (KSP inhibitor) are associated with toxicity and clinical outcome in patients with colorectal cancer. Further, whether genes involved with the metabolism (CYP3A4) and resistance (MDR1) affect the outcome in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive SB-715992 IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive SB-715992 IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced/metastatic colorectal cancer
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Patients must have received prior therapy (in any setting) with 5-FU, CPT-11, and oxaliplatin; patients may have received prior erbitux and bevacizumab, but it is not required
* Patients must have received at least one prior chemotherapy regimen for advanced disease
* Tumor must be accessible for biopsy or paraffin embedded tissue must be available for review of their biopsy specimen
* Life expectancy of > 12 weeks
* ECOG performance status 0-2 (Karnofsky >= 50%)
* Leukocytes >= 3,000/μL
* Absolute neutrophil count >= 1,500/μL
* Platelets >= 100,000/μL
* Hemoglobin >= 9 mg/dL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine =< 1.5 X institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from AEs due to agents administered more than 4 weeks earlier
* Patients may not have received any other investigational agents within 28 days of study entry
* Patients may not receive other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) while on this study
* Prohibited medications; SB-715992 is a moderate to significant in vitro inhibitor of CYP3A4; the following lists of medications/substances are moderate to significant inhibitors/inducers of CYP3A4 that, if administered concomitantly with SB-715992, may alter study drug exposure; the use of these medications/substances within 14 days (> 6 months for amiodarone) prior to the administration of the first dose of SB-715992 through discontinuation from the study is prohibited

  * Inhibitors of CYP3A4:

    * Antibiotics: clarithromycin, erythromycin, troleandomycin
    * Antifungals: itraconazole, ketoconazole, fluconazole (doses > 200 mg/day), voriconazole
    * Antidepressants: nefazodone, fluovoxamine
    * Calcium channel blockers: verapamil, diltiazem
    * Miscellaneous: amiodarone*, grapefruit juice, bitter orange

      * Use of amiodarone within 6 months prior to the administration of the first dose of SB-715992 is prohibited
  * Inducers of CYP3A4:

    * Anticonvulsants: phenytoin, carbamazepine, Phenobarbital, oxcarbazepine
    * Antibiotics: rifampin, rifabutin, rifapentine
    * Miscellaneous: St. John's wort, modafinil
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SB-715992
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with SB-715992
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-01; Primary Completion 2010-01 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, MD, Principal Investigator — University of Southern California, Norris
Locations (1):
- University of Southern California, Norris, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients receive SB-715992 IV at 7 mg/m2 over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  ispinesib: Given IV
  laboratory biomarker analysis: Correlative studies
- Arm II: Patients receive SB-715992 IV at 18 mg/m2 over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  ispinesib: Given IV
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 33 | 31
Completed | 29 | 30
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Median (Full Range); unit: years] | 59 [28 to 82] | 60 [35 to 80] | 59 [28 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 19 | 18 | 37
Region of Enrollment [Number; unit: participants]
  United States | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (CR or PR) as Determined by the RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 33 | 31
participants | 0 | 0

2. Secondary Outcome: Progression-free Survival
Description: Will be estimated using the product-limit method of Kaplan and Meier by arm. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the date of registration to the date of documented PSA progression, assessed up to 6 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 33 | 31
weeks | 7.0 [6.3 to 7.3] | 5.3 [5.0 to 5.9]

3. Secondary Outcome: Overall Survival
Description: Will be estimated using the product-limit method of Kaplan and Meier by arm.
Time Frame: From the date of registration to the date of death, assessed up to 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 33 | 31
months | 3.6 [2.5 to 8.2] | 4.5 [3.7 to 7.0]

ADVERSE EVENTS:
Time Frame: Adverse events were over a period of 4 years.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 14/33 | 13/31
Other Adverse Events (participants affected / at risk) | 33/33 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=33) | Arm II (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 2 (2)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Hyperbilirubinemia (Investigations) | 1 (1) | 3 (3)
INR increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 8 (8)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=33) | Arm II (N=31)
Hemoglobin decreased (Blood and lymphatic system disorders) | 17 (23) | 18 (29)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Flashing vision (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 14 (21) | 10 (12)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (13) | 10 (14)
Diarrhea (Gastrointestinal disorders) | 8 (10) | 8 (10)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (12) | 10 (13)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (7) | 8 (8)
Disease progression (General disorders) | 29 (29) | 24 (24)
Edema limbs (General disorders) | 4 (5) | 4 (6)
Fatigue (General disorders) | 20 (40) | 19 (29)
Fever (General disorders) | 2 (3) | 5 (5)
Localized edema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 8 (10) | 3 (4)
Alkaline phosphatase increased (Investigations) | 13 (24) | 16 (28)
Aspartate aminotransferase increased (Investigations) | 13 (19) | 13 (23)
Cardiac troponin T increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 1 (1)
Hyperbilirubinemia (Investigations) | 8 (10) | 4 (4)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1)
Leukopenia (Investigations) | 6 (8) | 13 (17)
Lymphopenia (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 9 (12) | 15 (19)
Platelet count decreased (Investigations) | 2 (3) | 7 (9)
Weight loss (Investigations) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 13 (22) | 11 (16)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (15) | 10 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (12) | 10 (15)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 7 (9)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 5 (11) | 7 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (9) | 9 (16)
Agitation (Psychiatric disorders) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 4 (5) | 5 (8)
Confusion (Psychiatric disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 3 (4) | 5 (6)
Euphoria (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 9 (10)
Personality change (Psychiatric disorders) | 1 (2) | 0 (0)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (4)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (7) | 5 (9)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 5 (8) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 2 (2) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less